CLINICAL TRIAL: NCT06667635
Title: Intelligent Analysis and Clinical Validation of Cerebral Small Vessel Disease on Magnetic Resonance Imaging：A Multi-center Study
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: 2024-685
Record Dates: First submitted 2024-10-22; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Small Vessel Disease
Keywords: Cerebral small vessel disease; Artificial intelligence; Deep learning; Magnetic resonance imaging
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Artificial intelligence — Artificial intelligence (AI) tools developed through the training of large amounts of image data can assist with the analysis and interpretation of neuroimaging data of cerebral small vascular disease（CSVD）.

SUMMARY:
Cerebral small vessel disease (CSVD) accounts for 20% of ischemic strokes and is the most common cause of vascular cognitive impairment. Early identification of CSVD is critical for early intervention and improve clinical outcomes. Magnetic resonance imaging (MRI) may represent as a sensitive and robust tool to detect early changes in brain subtle structures and functions. The study is to investigate the comprehensive evaluation by using AI in early diagnosis and management of CSVD.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) is an important cause of stroke, cognitive impairment, and other diseases, and its early quantitative evaluation can significantly improve patient prognosis. Magnetic resonance imaging (MRI) is an important method to evaluate the occurrence, development, and severity of CSVD. However, the diagnostic process lacks quantitative evaluation criteria and is limited by experience, which may easily lead to missed diagnoses and misdiagnoses. Based on the current technical challenges, subject development and upgrade of knowledge, to avoid the occurrence of adverse medical accidents, simplify the diagnostic process, artificial intelligence（AI） has become the alternative method of choice, by constructing training deep learning model,which can assist doctors in clinical decision-making to improve diagnosis effectiveness of CSCD detection and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* ① Men and women age 40 years or older;

  * At least one vascular risk factor has been identified, including hypertension, diabetes, hyperlipidemia, coronary heart disease, and chronic kidney disease；

    * The patient performed two brain MRI Examinations simultaneously at a time interval of more than 6 months (≥6).

Exclusion Criteria:

* ① The patient had no vascular risk factors；

  * No clinical follow-up images;

    * There are significant motion artifacts in the image, which cannot meet the

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a multicenter study with a total plan of 1000 patients, 500 from Chinese PLA General Hospital and 500 from other centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
The performance of AI in lesion detection and diagnosis | 2 year
  The performance of AI in lesion detection and diagnosis, including imaging quality, accuracy, sensitivity and specificity in lesion detection and imaging diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD/PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China, China